CLINICAL TRIAL: NCT03948217
Title: The Effects of Artificial Lighting on Affective and Core Symptoms of Eating Disorder - a Pilot Study
Brief Title: The Effects of Artificial Lighting on Affective and Core Symptoms of Eating Disorder
Acronym: METROPOLIS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: changes to buildings why study was terminated prematurely
Sponsor: Mental Health Centre Copenhagen, Bispebjerg and Frederiksberg Hospital (Other)
Collaborators: Aalborg University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: H-17022914
Record Dates: First submitted 2019-05-03; First posted 2019-05-13 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Anorexia Nervosa; Eating Disorder
Keywords: artificial lighting
MeSH Terms: conditions — Anorexia Nervosa; Feeding and Eating Disorders

STUDY DESIGN:
Intervention Model Description: Single blind, cross-over, controlled
Who Masked: Participant, Care Provider
Masking Description: Patients are unaware of the type of Circadian lighting regimen that is provided
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- L1 (Active Comparator): regimen L1 has overall higher intensity, higher color temperature and less light fluctuations
  Interventions: Other: Circadian Lighting regimen
- L2 (Active Comparator): regimen L2 has lower intensity, lower color temperature and more light fluctuations.
  Interventions: Other: Circadian Lighting regimen

INTERVENTIONS:
Other: Circadian Lighting regimen — Circadian lighting regimen with one major fluctuation, high light intensity and color

SUMMARY:
The primary objective of this pilot study is to explore the effect of artificial lighting on affective symptoms, and the secondary aim is to explore the effect of artificial lighting on core symptoms of eating disorders (ED).

Several lines of evidence, albeit from hypothesis generation studies, suggest that artificial lighting may have a positive effect on well-being, mental health and affective symptoms in ED. The rationale of this study is to investigate the effects of artificial lighting on affective symptoms and cores symptoms of ED in inpatients undergoing weight restoration/treatment for ED.

Study design: Single-blind, controlled, pilot intervention study with circadian light (CL) comparing two CL regimens effects on mood symptoms.

Planned number of subjects: 16 patients with a ICD-10 diagnosis of Anorexia Nervosa, that completes exposure to at least three weeks of the two different CL regimens (L1 and L2) in any order.

DETAILED DESCRIPTION:
The primary objective of this pilot study is to explore the effect of artificial lighting on affective symptoms, and the secondary aim is to explore the effect of artificial lighting on core symptoms of eating disorders (ED).

If an effect is indicated, the study will provide information on how to improve light exposure to ED patients in psychiatric treatment units. In addition, the outcomes may help identify a better system for measurement and adjustment of the specific light variables of colour temperature and light intensity.

Several lines of evidence, albeit from hypothesis generation studies, suggest that artificial lighting may have a positive effect on well-being, mental health and affective symptoms in ED. This is the rationale to investigate the effects of artificial lighting on affective symptoms and cores symptoms of ED in inpatients undergoing weight restoration/treatment for ED.

Study design: Single-blind, controlled, pilot intervention study with circadian light (CL) comparing two CL regimens effects on mood symptoms.

Planned number of subjects: 16 patients with a International Classification of Disorders 10 (ICD-10) diagnosis of Anorexia Nervosa, that completes exposure to at least three weeks of the two different CL regimens (L1 and L2) in any order.

Location: Mental Health Center Ballerup, department 14 (currently Department 5).

Diagnostic inventory: Eating Disorder Examination-Questionnaire (EDE-Q)

ELIGIBILITY:
Inclusion Criteria:

1. Primary diagnosis of Anorexia Nervosa (AN) or Bulimia Nervosa (BN) or Eating Disorder Not Otherwise specified (EDNOS)
2. Age ≥18 and <65

Exclusion Criteria:

1. Forced care
2. Non-primary psychiatric disorder other than AN, BN, or EDNOS
3. Binge Eating disorder
4. Somatic unstable condition
5. High suicidal behavior or risk

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2018-07-31 (Actual); Study Completion 2018-08-31 (Actual)

PRIMARY OUTCOMES:
3 week change in total score of Major Depression Inventory | 3 weeks change from baseline
  depression scoring, change in total score over three weeks. range 0-50. Higher values means more depressed. Mild depression: MDI total score from 21 to 25. Moderate depression: MDI total score from 26 to 30. Severe depression: MDI total score of 31 or higher.
3 week change in total score of Eating Disorder Inventory 2 | 3 weeks change from baseline
  Eating disorder symptoms total score change over 3 weeks. range 0-273. Higher score means more Eating disorder symptoms.
3 week change in video images based measure of Physical activity | 3 weeks change in physical activity from baseline
  video images based measure of quantity of physical activity

SECONDARY OUTCOMES:
3 week change in BMI | 3 week change as a measure of weight change
  change in Body Mass index
3 week change in Visual analogue scale of mood | 3 weeks change from baseline
  self assessed measure of mood symptoms, range 1-10. Higher score means more symptoms and feeling worse.
3 week change in melatonin levels | 3 weeks change from baseline
  urinary levels of melatonin
3 week change in serotonin levels | 3 weeks change from baseline
  Blood levels of serotonin
3 week change in cortisol levels | 3 weeks change from baseline
  Urinary levels of cortisol as a measure of stress

CONTACTS AND LOCATIONS:
Locations (1):
- Mental Health Center, Ballerup Municipality, Capitol Region, Denmark

IPD SHARING:
Plan to Share IPD: Yes
All patient data
Supporting Information: Study Protocol
Time Frame: within 12 months
Access Criteria: open